CLINICAL TRIAL: NCT06999018
Title: Humeral Shaft Fractures : Outcomes of Straight Percutaneous Intramedullary Nailing With Dynamic Distal Locking
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0013_HUMERUS
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: COVID-19; Coronavirus Infections; Seroprevalence; Vaccination; Health Care Workers
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study looks at how many healthcare workers at CHSD have developed antibodies against COVID-19 after the second and third waves of the pandemic and following vaccination. By testing blood samples, we want to understand how well healthcare workers are protected, which work areas might be more at risk, and how immunity changes over time after infection or vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated between January 2008 and June 2018
* Closed, isolated, displaced fractures of the humeral shaft
* Treatment by percutaneous anterograde intramedullary nailing with dynamic distal locking
* Availability for follow-up and evaluation (e.g., Constant score assessment in June 2018)

Exclusion Criteria:

* Open fractures
* Fractures that are not isolated or not displaced
* Patients lost to follow-up at the June 2018 evaluation (18 excluded)
* Lack of Constant score evaluation (patients not reviewed)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult patients who underwent surgical treatment for closed, isolated, and displaced fractures of the humeral shaft. These patients were treated with percutaneous anterograde intramedullary nailing using dynamic distal locking between January 2008 and June 2018. The population includes both men and women, with a mean age of approximately 53 years. Only patients with fractures classified as type A, B, or C according to the AO/OTA classification and who were available for follow-up evaluation were included. Patients with open fractures, non-isolated or non-displaced fractures, or those lost to follow-up were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The seroprevalence of SARS-CoV-2 antibodies among healthcare workers at CHSD following COVID-19 vaccination and previous infection. | January 2008 - June 2018

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France